CLINICAL TRIAL: NCT00113568
Title: Multicenter Study to Evaluate the Safety of XP12B in Women With Heavy Menstrual Bleeding Associated With Menorrhagia
Brief Title: Safety Study of XP12B in Women With Menorrhagia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XP12B-MR-302
Record Dates: First submitted 2005-06-08; First posted 2005-06-09 (Estimated); Results first posted 2010-01-20 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2010-06

CONDITIONS: Menorrhagia; Heavy Menstrual Bleeding
Keywords: Menorrhagia; Heavy Menstrual Bleeding
MeSH Terms: conditions — Menorrhagia | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- XP12B (tranexamic acid tablets) (Experimental)
  Interventions: Drug: Tranexamic acid tablets (XP12B)

INTERVENTIONS:
Drug: Tranexamic acid tablets (XP12B) — Two 650 mg tranexamic acid tablets (XP12B) taken 3 times daily (3900 mg/Day) for a maximum of 5 days during monthly menstruation
  Other Names: Lysteda; XP12B; tranexamic acid tablets; XP12B-MR

SUMMARY:
The purpose of this study is to evaluate the safety of XP12B in women with heavy menstrual bleeding associated with menorrhagia.

ELIGIBILITY:
Inclusion Criteria:

* Women with menorrhagia
* 18-49 years of age
* Regularly occuring menstrual periods

Exclusion Criteria:

* History or presence of clinically significant disease or abnormalities that might confound the study
* History of bilateral oophorectomy or hysterectomy

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 784 (Actual)
Dates: Start 2005-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (50):
- United States (50):
  - Investigative Site, Birmingham, Alabama
  - Investigative Site, Mobile, Alabama
  - Investigative Site, Montgomery, Alabama
  - Investigative Site, Phoenix, Arizona
  - Investigative Site, Jonesboro, Arkansas
  - Investigative Site, Little Rock, Arkansas
  - Investigative Site, San Diego, California
  - Investigative Site, Colorado Springs, Colorado
  - Investigative Site, Denver, Colorado
  - Investigative Site, Fort Myers, Florida
  - Investigative Site, Miami, Florida
  - Investigative Site, New Port Richey, Florida
  - Investigative Site, Ocala, Florida
  - Investigative Site, Pinellas Park, Florida
  - Investigative Site, Venice, Florida
  - Investigative Site, West Palm Beach, Florida
  - Investigative Site, Alpharetta, Georgia
  - Investigative Site, Roswell, Georgia
  - Investigative Site, Savannah, Georgia
  - Investigative Site, Boise, Idaho
  - Investigative Site, Champaign, Illinois
  - Investigative Site, Evansville, Indiana
  - Investigative Site, Indianapolis, Indiana
  - Investigative Site, South Bend, Indiana
  - Investigative Site, Overland Park, Kansas
  - Investigative Site, Lexington, Kentucky
  - Investigative Site, Louisville, Kentucky
  - Investigative Site, Shreveport, Louisiana
  - Investigative Site, Portage, Michigan
  - Investigative Site, Chaska, Minnesota
  - Investigative Site, St Louis, Missouri
  - Investigative Site, Billings, Montana
  - Investigative Site, Omaha, Nebraska
  - Investigative Site, Las Vegas, Nevada
  - Investigative Site, Moorestown, New Jersey
  - Investigative Site, Albuquerque, New Mexico
  - Investigative Site, Johnson City, New York
  - Investigative Site, Charlotte, North Carolina
  - Investigative Site, Durham, North Carolina
  - Investigative Site, Winston-Salem, North Carolina
  - Investigative Site, Cincinnati, Ohio
  - Investigative Site, Toledo, Ohio
  - Investigative Site, Philadelphia, Pennsylvania
  - Investigative Site, Wexford, Pennsylvania
  - Investigative Site, Columbia, South Carolina
  - Investigative Site, Nashville, Tennessee
  - Investigative Site, Houston, Texas
  - Investigative Site, Norfolk, Virginia
  - Investigative Site, Seattle, Washington
  - Investigative Site, Tacoma, Washington

REFERENCES:
- [Derived] Muse K, Lukes AS, Gersten J, Waldbaum A, Mabey RG, Trott E. Long-term evaluation of safety and health-related quality of life in women with heavy menstrual bleeding treated with oral tranexamic acid. Womens Health (Lond). 2011 Nov;7(6):699-707. doi: 10.2217/whe.11.65. Epub 2011 Aug 25. PMID 21867401
- [Derived] Bushnell DM, Martin ML, Moore KA, Richter HE, Rubin A, Patrick DL. Menorrhagia Impact Questionnaire: assessing the influence of heavy menstrual bleeding on quality of life. Curr Med Res Opin. 2010 Dec;26(12):2745-55. doi: 10.1185/03007995.2010.532200. Epub 2010 Nov 3. PMID 21043553

RESULTS

PARTICIPANT FLOW:
Groups:
- Tranexamic Acid Tablets (XP12B): Two 650 mg tranexamic acid tablets taken 3 times daily (3900 mg/day) for a maximum of 5 days during monthly menstruation
Period: Overall Study
Arm/Group | Tranexamic Acid Tablets (XP12B)
Started | 784
Intent to Treat Population | 723
Completed | 239
Not Completed | 545
Not completed — Adverse Event | 97
Not completed — Death | 1
Not completed — Lack of Efficacy | 30
Not completed — Lost to Follow-up | 156
Not completed — Protocol Violation | 32
Not completed — Withdrawal by Subject | 117
Not completed — Other | 112

BASELINE CHARACTERISTICS:
Arm/Group | Tranexamic Acid Tablets (XP12B)
Number analyzed (Participants) | 723
Age Continuous [Mean (Standard Deviation); unit: years] | 38 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 723
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Adverse Event During the Study
Description: An adverse event is any untoward, undesired, unplanned clinical event in the form of signs. symptoms, disease, or laboratory or physiological observations occurring in a human being participating in a clinical study with a sponsor study drug, regardless of causal relationship.
Time Frame: Up to 27 menstrual cycles
Population: intent to treat population
Measure: Number; unit: participants
Arm/Group | Tranexamic Acid Tablets (XP12B)
Number analyzed (Participants) | 723
participants | 678

2. Primary Outcome: Number of Subjects With at Least One Possibly Treatment-Related Adverse Event During the Study
Description: The causal relation between an adverse event and the study drug was determined by the investigator on the basis of his or her clinical judgment. A possibly treatment-related adverse event is an event that may be explained by administration of the study drug or by the subjects's clinical state or other agents/therapies.
Time Frame: Up to 27 menstrual cycles
Population: intent to treat population
Measure: Number; unit: participants
Arm/Group | Tranexamic Acid Tablets (XP12B)
Number analyzed (Participants) | 723
participants | 306

3. Primary Outcome: Number of Subjects With at Least One Probably Treatment-Related Adverse Event During the Study
Description: The causal relation between an adverse event and the study drug was determined by the investigator on the basis of his or her clinical judgment. A probably treatment-related adverse event is an event most likely to be explained by administration of the study drug rather than the subjects's clinical state or other agents/therapies.
Time Frame: Up to 27 menstrual cycles
Population: intent to treat population
Measure: Number; unit: participants
Arm/Group | Tranexamic Acid Tablets (XP12B)
Number analyzed (Participants) | 723
participants | 40

4. Primary Outcome: Number of Subjects With at Least One Definitely Treatment-Related Adverse Event During the Study
Description: The causal relation between an adverse event and the study drug was determined by the investigator on the basis of his or her clinical judgment. A definitely treatment-related adverse event is an event that can be fully explained by administration of the study drug.
Time Frame: Up to 27 menstrual cycles
Population: intent to treat population
Measure: Number; unit: participants
Arm/Group | Tranexamic Acid Tablets (XP12B)
Number analyzed (Participants) | 723
participants | 13

5. Primary Outcome: Number of Subjects With at Least One Serious Adverse Event During the Study
Description: A serious adverse event (SAE) is any adverse event (AE) occurring at any dose that meets 1 or more of the following criteria: results in death; is life-threatening; requires inpatient hospitalization or prolongation of an existing hospitalization; results in a persistent or significant disability or incapacity; results in cancer; results in a congenital anomaly or birth defect. Important medical events not described above may be considered SAEs when based on appropriate medical judgment.
Time Frame: Up to 27 menstrual cycles
Population: intent to treat population
Measure: Number; unit: participants
Arm/Group | Tranexamic Acid Tablets (XP12B)
Number analyzed (Participants) | 723
participants | 28

6. Primary Outcome: Number of Subjects With at Least One Life-Threatening Adverse Event During the Study
Description: A life-threatening AE is any AE that places the subject at immediate risk of death from the event as it occurred.
Time Frame: Up to 27 menstrual cycles
Population: intent to treat population
Measure: Number; unit: participants
Arm/Group | Tranexamic Acid Tablets (XP12B)
Number analyzed (Participants) | 723
participants | 2

7. Primary Outcome: Number of Subjects With Adverse Events That Led to Discontinuation From the Study
Description: The total number of subjects who withdrew from the study due to an adverse event irrespective of the causal relation between the AE and the study drug as determined by the investigator
Time Frame: Up to 27 menstrual cycles
Measure: Number; unit: participants
Arm/Group | Tranexamic Acid Tablets (XP12B)
Number analyzed (Participants) | 784
participants | 97

8. Primary Outcome: Number of Subjects With Any Thrombotic or Thromboembolic Adverse Event During the Study
Description: Examples include deep vein thrombosis, pulmonary embolism, cerebral thrombosis, acute renal cortical necrosis, central retinal artery and vein obstruction.
Time Frame: Up to 27 menstrual cycles
Population: intent to treat population
Measure: Number; unit: participants
Arm/Group | Tranexamic Acid Tablets (XP12B)
Number analyzed (Participants) | 723
participants | 0

9. Primary Outcome: Number of Subjects Who Died During the Study
Description: Number of subjects who died, for any reason, during the study
Time Frame: Up to 27 menstrual cycles
Measure: Number; unit: participants
Arm/Group | Tranexamic Acid Tablets (XP12B)
Number analyzed (Participants) | 784
participants | 1

ADVERSE EVENTS:
Arm/Group | Tranexamic Acid Tablets (XP12B)
Serious Adverse Events (participants affected / at risk) | 28/723
Other Adverse Events (participants affected / at risk) | 678/723
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tranexamic Acid Tablets (XP12B) (N=723)
Anemia (Blood and lymphatic system disorders) | 1
Cardiac Arrest (Cardiac disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Hiatus Hernia (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Abdominal Wall Abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Glycopeptide antiobiotic resistant staphylococcal aureus infection (Infections and infestations) | 1
Malaria (Infections and infestations) | 1
Aseptic meningitis (Infections and infestations) | 1
Pneumococcal sepsis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Wound Abscess (Infections and infestations) | 1
Animal Bite (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 2
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 4
Neuritis (Nervous system disorders) | 1
Partial seizures with secondary generalization (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Depression (Psychiatric disorders) | 1
Adenomyosis (Reproductive system and breast disorders) | 1
Dysmenorrhea (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 4
Uterine Leiomyoma (Reproductive system and breast disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tranexamic Acid Tablets (XP12B) (N=723)
Anemia (Blood and lymphatic system disorders) | 37
Abdominal Discomfort (Gastrointestinal disorders) | 87
Upper abdominal pain (Gastrointestinal disorders) | 65
Diarrhea (Gastrointestinal disorders) | 88
Dyspepsia (Gastrointestinal disorders) | 60
Nausea (Gastrointestinal disorders) | 104
Toothache (Gastrointestinal disorders) | 42
Vomiting (Gastrointestinal disorders) | 43
Fatigue (General disorders) | 57
Multiple allergies (Immune system disorders) | 39
Seasonal allergy (Immune system disorders) | 66
Sinusitis (Infections and infestations) | 94
Upper respiratory tract infection (Infections and infestations) | 68
Urinary tract infection (Infections and infestations) | 45
Viral upper respiratory tract infection (Infections and infestations) | 137
Post procedural pain (Injury, poisoning and procedural complications) | 51
Arthralgia (Musculoskeletal and connective tissue disorders) | 105
Back pain (Musculoskeletal and connective tissue disorders) | 227
Muscle cramp (Musculoskeletal and connective tissue disorders) | 41
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 98
Myalgia (Musculoskeletal and connective tissue disorders) | 50
Neck pain (Musculoskeletal and connective tissue disorders) | 61
Pain in extremity (Musculoskeletal and connective tissue disorders) | 100
Dizziness (Nervous system disorders) | 50
Headache (Nervous system disorders) | 437
Migraine (Nervous system disorders) | 78
Sinus headache (Nervous system disorders) | 70
Insomnia (Psychiatric disorders) | 74
Dysmenorrhea (Reproductive system and breast disorders) | 78
Menstrual discomfort (Reproductive system and breast disorders) | 360
Cough (Respiratory, thoracic and mediastinal disorders) | 80
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 64
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 69
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 100
Menorrhagia (Reproductive system and breast disorders) | 40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other